CLINICAL TRIAL: NCT02913014
Title: Monitoring Safety and Recurrence of Paroxysmal Atrial Fibrillation After 1st Cryo-balloon Ablation with and Without Antiarrhythmic Drug Therapy During the 90-day Blanking Period - Examined with Adverse Event Monitoring and Cardiovascular Implantable Electronic Devices (CIEDs)
Brief Title: Comparison of Recurrence of Atrial Fibrillation Post Cryoballon Ablation During the 90-day Blanking Period-with and Without Anti-arrhythmic Drug Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Midlands (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00055684
Record Dates: First submitted 2016-08-31; First posted 2016-09-23 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: Antiarrhythmic Agents; Catheter Ablation, electric; Cardiac Arrhythmias; Anti-Arrhythmia Drugs
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1- No AAD post Ablation (Active Comparator): Subjects will not resume their Anti Arrhythmic Drugs after cryoballoon-ablation for paroxysmal atrial fibrillation.
  Interventions: Other: No AAD post Ablation.
- Arm 2-Resume AAD post Ablation (No Intervention): Subjects will resume their pre-ablation Anti Arrhythmic Drugs after cryoballoon-ablation for paroxysmal atrial fibrillation, during the 90 day blanking period following the ablation.

INTERVENTIONS:
Other: No AAD post Ablation. — Subjects will not resume their pre-ablation anti-arrhythmic medications during the 90 following cryo ablation for Atrial Fibrillation
  Other Names: No AAD
  Arms: Arm 1- No AAD post Ablation

SUMMARY:
This study is being done to find out if patients taking Anti Arrhythmia Drugs (AADs) after cryoballoon ablation for atrial fibrillation, compared to patients who do not take Anti- Arrhythmic Drugs after an ablation affect Atrial Fibrillation from coming back. The study will also look at the side effects of the AADs.

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) is a cornerstone ablation strategy used in the management of paroxysmal atrial fibrillation (PAF), and it is a class IA indication for anti-arrhythmic drug (AAD) refractory symptomatic PAF. However, the consensus statements are vague about the utility of AAD management during the 90-day blanking window post-PVI. Moreover, there is no specific guidance to cryoballoon users on the usage of AADs during the 90-day blanking period that exists anywhere in the published literature. Simply, these studies have not been conducted with the cryoballoon procedure.

ELIGIBILITY:
Inclusion Criteria:

* Drug refractory and recurrent Paroxysmal Atrial Fibrillation
* The subject meets medical criteria for cryoballoon ablation to treat Paroxysmal AF
* Age 18 to 80 years
* The subject has a Cardiovascular Implantable Electronic Device (CIED) that captures AF episodes, such as an implantable loop recorder, pacemaker, or implantable cardioverter defibrillator (ICD) with a properly functioning atrial lead.

Exclusion Criteria:

* Use of any Anti- Arrhythmic Drugs for ventricular arrhythmias
* Ejection Fraction (EF)<45%
* Prior A. Fib. ablation
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Compare recurrence, recurrence rate, burden of atrial fibrillation post ablation between the two groups. | 12 months
  Rhythm status through implantable loop recorder (or pacemaker with functioning atrial lead) at 3 month, 6 month, 12 month compared between two treatment groups, including:
  A) AF burden (Average amount of time in AF per day) B) AF recurrence rate (Frequency of AF, occurrences per day) C) Time to AF recurrence
Symptom Assessments | 12 months
  Symptom assessments by clinical follow up and phone calls, including symptom severity score using the Severity of Atrial Fibrillation Scale between the two groups.
Adverse Events Assessments | 12 months
  Ongoing assessment of adverse events in both arms of the study, including AADs side effects in 90-day blanking period.

SECONDARY OUTCOMES:
The cost of AADs during the 90-day blanking period. | 12 months
  The cost of AADs during the 90-day blanking period.
Assess the rate of hospitalizations, emergency room visits, and unscheduled cardiology visits for the treatment of AF between the two groups | 12 months
  A) Event during the 90-day blanking period will be assessed for AAD related and unrelated adverse events that caused the cardiac related visit
The differential usage of anticoagulation therapy between two arms. | 12 months
  The differential usage of anticoagulation therapy between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan M Siddique, MD, Principal Investigator — Prisma Health-Midlands
Locations (1):
- Palmetto Health, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No